CLINICAL TRIAL: NCT06472778
Title: Smoldering Pathway Assessment Real-World Knowledge (SPARK) Study-Retrospective Observational, Non-interventional Chart Review Study in Smoldering Multiple Myeloma
Brief Title: A Real-world Study in Participants With Smoldering Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 54767414SMM4001; 54767414SMM4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Participants with Smoldering Multiple Myeloma (SMM): Participants diagnosed with SMM between 01 January 2016 and 31 December 2021 will be enrolled in this study. Only data available outside of clinical studies from participant medical records will be collected. The data collected per participant in this study is defined as data available in medical charts from date of SMM diagnosis until 31 December 2023, death or lost to follow-up, whichever comes first.

SUMMARY:
The purpose of this study is to evaluate the real-world characteristics and outcomes of participants with smoldering multiple myeloma (SMM) overall and by high-risk and non-high-risk SMM according to (AQUILA study criteria [NCT03301220], Mayo 20-2-20 and international myeloma working group (IMWG) 2020 risk classification models), and to evaluate the risk of progressing of SMM to multiple myeloma (MM) and outcomes in participants after progressing to MM.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of smoldering multiple myeloma (SMM). SMM is defined as: (a) Clonal bone marrow plasma cells (BMPCs) greater than or equal to (>=) 10 percent (%) and/or serum M-protein >= 3 grams per deciliter (g/dL) and/or urine M-protein >= 500 milligram per 24 hours (mg/24hrs). (b) Absence of SLiM-CRAB criteria: >= 60 % clonal BMPCs, involved/uninvolved free light chain (FLC) ratio >= 100 and involved FLC >= 10 and magnetic resonance imaging (MRI) lesions; calcium elevation, renal insufficiency, anemia, and bone lesions (AB) criteria
* Informed consent obtained prior to retrospective data collection in accordance with local requirements, either an informed consent form (ICF) indicating that the participants signed a consent for data collection for this research and agrees to have their data collected and analyzed, with source data verification (SDV), or the country does accept the ICF waiver for such type of studies
* Data recorded in participants' medical charts from date of SMM diagnosis and at least 2 years after should be available in the participant's medical chart at the participating site. However, participants who died within the 2 years from SMM diagnosis are eligible

Exclusion Criteria:

* Therapy for multiple myeloma (MM) initiated within 90 days of SMM diagnosis
* Date of SMM diagnosis is missing
* Participants who have participated/are participating in any SMM interventional (either active treatment or control arm) study are not eligible. Participation in observational studies is allowed. Participants who have participated/are participating in any MM study after evolution to MM are eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants aged at least 18 years of age on the date of documented diagnosis of smoldering multiple myeloma (SMM) between 01 January 2016 and 31 December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Participant Characteristics and Treatment Patterns: Number of Participants With Type of Treatment | Data collection up to 1 year and 2 months
  Number of participants with type of treatment (example, autologous stem cell transplant [ASCT], chimeric antigen receptor [CAR-T], proteasome inhibitor [PI], and immunomodulatory drug [iMID]) will be reported in participants with smoldering multiple myeloma (SMM) overall and by high-risk and non-high-risk classifications.
Participant Characteristics and Treatment Patterns: Duration of Treatment | Data collection up to 1 year and 2 months
  Duration of treatment as defined from the date of first dose of SMM treatment until the last dose of SMM treatment by treatment type will be reported.
Participant Characteristics and Treatment Patterns: Time to Best Response | Data collection up to 1 year and 2 months
  Time to best response is defined as the time interval from the date of first dose of SMM treatment until recorded best response, by treatment type. Time to best response for SMM treatments will not be collected for countries which do not allow it.
Participant Characteristics and Treatment Patterns: Overall Survival in Participants With SMM Overall and for High-risk and Non-high-risk Participants | Data collection up to 1 year and 2 months
  Overall survival is defined as the time interval from the date of SMM diagnosis until the date of last observation (that is, date of end of study for each participant) or death, whichever comes first.
Observation Patterns for High-risk and Non-high-risk SMM Participants and Overall | Data collection up to 1 year and 2 months
  Observational patterns (example, frequency of visits and hospitalizations) will be reported for high-risk and non-high-risk SMM participants and overall.
Time to Progression to Multiple Myeloma (MM) in Participants With High-risk SMM | Data collection up to 1 year and 2 months
  Time to progression to multiple myeloma (MM) is defined as the the time from the date of SMM diagnosis to the date of MM diagnosis, as defined by 60 percent plasma cells, light chains, and MRI lesions (SLiM) and/or calcium elevation, renal insufficiency, anemia, and bone lesions (CRAB) criteria.
Progression-free Survival | Data collection up to 1 year and 2 months
  Progression-free survival defined from the date of SMM diagnosis until date of MM diagnosis or death of any cause, whichever occurs first.
Rates of Progression From SMM to MM for High and Non-high-risk Participants | Data collection up to 1 year and 2 months
  Rate of progression from SMM to MM for high and non-high-risk participants will be evaluated as per SliM and/or CRAB criteria.
Risk Factors of Progression From SMM to MM | Data collection up to 1 year and 2 months
  Potential risk factors/predictors for progression from SMM diagnosis to MM will be investigated, for high-risk participants and non-high-risk participants according to AQUILA study criteria (NCT03301220), Mayo 20-2-20 and international myeloma working group (IMWG) 2020 risk stratification models, example age at SMM diagnosis and eastern cooperative oncology group (ECOG) at SMM diagnosis.
Number of Participants With Myeloma-related Organ Damage Who Progress From SMM to MM | Data collection up to 1 year and 2 months
  Number of participants with outcomes of myeloma-related organ damage who progress from SMM to MM will be summarized overall and by high-risk and non-high-risk participants.

SECONDARY OUTCOMES:
Percentage of Participants With High-risk and Non-high-risk SMM | Baseline
  Percentage of participants with high-risk and non-high-risk SMM will be reported.
Participant Characteristics With High-risk and Non-high-risk SMM | Data collection up to 1 year and 2 months
  Participant characteristics with high-risk and non-high risk SMM (example, age at SMM and MM diagnosis, date of SMM and MM diagnosis, Sex at birth, ECOG, and country) will be reported.
Best Response for the First-Line Treatment for MM | Data collection up to 1 year and 2 months
  Best Response on first-line MM therapy (stringent complete response [sCR], complete response [CR], and partial response [PR]) will be reported based on the IMWG response criteria. Best response for SMM treatments will not be collected for countries which do not allow it.
Time to Best Response to MM Treatment | Data collection up to 1 year and 2 months
  Time to best response to MM treatment defined as the time interval from the date of first dose of MM treatment until recorded best response, by treatment type. Time to best response for SMM treatments will not be collected for countries which do not allow it.
Number of Participants with Type of MM Treatment | Data collection up to 1 year and 2 months
  Number of participants with type of MM treatment will be reported for participants whose SMM evolved to MM.
Duration of MM Treatment | Data collection up to 1 year and 2 months
  Duration of treatment defined from the date of first dose for MM until the last dose of MM treatment, by type of treatment will be reported.
Overall Survival for Participants Whose SMM Evolved to MM | Data collection up to 1 year and 2 months
  Overall survival is defined as the time interval from the date of SMM diagnosis until the date of last observation (that is, date of end of study for each participant) or death, whichever comes first.
Disease Progression Related Deaths | Data collection up to 1 year and 2 months
  Disease progression related deaths will be reported. Disease progression related deaths defined as the time from the date of SMM diagnosis to the date of death due to disease progression (primary cause).
Therapies Received | Data collection up to 1 year and 2 months
  Type, dose, and start/end date of relevant therapies received since SMM diagnosis will be reported.
Number of Participants With Adverse Drug Reactions (ADRs) | Data collection up to 1 year and 2 months
  Number of participants with ADRs as recorded in participants' medical charts will be reported.
Number of Participants With Abnormalities in Clinical Laboratory Tests | Data collection up to 1 year and 2 months
  Number of participants with abnormalities in clinical laboratory tests (only available hematology, chemistry, and bone marrow biopsy or aspirate results that are obtained as part of the participants' usual standard of care) will be reported.
Survival Status at End of Study | Data collection up to 1 year and 2 months
  Number of participants who were alive or dead at the end of the study will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (29):
- France (5):
  - CHRU de Tours - Hopital Trousseau, Chambray-lès-Tours
  - CHU Montpellier, Montpellier
  - Centre Hospitalier Regional d'Orleans (CHRO) - Hopital La Source, Orléans
  - Hopital Pitie Salpetriere, Paris
  - CH Rene Dubos, Pontoise
- Germany (4):
  - Studienzentrum Gefos Dortmund mbH, Dortmund
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - ELBLANDKLINIKUM Riesa, Riesa
  - Universitaetsklinikum Tuebingen, Tübingen
- Italy (5):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Universita di Roma La Sapienza, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino, Torino
- Spain (7):
  - Hosp Univ A Coruna, A Coruña
  - Hosp. Prov. de Avila, Ávila
  - Hosp. San Pedro de Alcantara, Cáceres
  - Hosp. Univ. Lucus Augusti, Lugo
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Clinico Univ. de Valladolid, Valladolid
  - Hosp. Univ. de Alava, Vitoria-Gasteiz
- United Kingdom (8):
  - Birmingham Heartlands Hospital, Birmingham
  - Kent and Canterbury Hospital, Canterbury
  - University Hospital of Wales, Cardiff
  - University Hospitals Of Leicester Nhs Trust, Leicester
  - Barts Hospital, London
  - Manchester Royal Infirmary, Manchester
  - South Tees Hospitals NHS Foundation Trust, North Yorks
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No